CLINICAL TRIAL: NCT07163169
Title: Correlation and Comparison Analyses of CARG, G8, and Frailty Tests in Predicting Chemotherapy-Associated Toxicity: A Prospective Study
Brief Title: Predicting Chemo Toxicity Using Geriatric Forms
Status: Active, not recruiting | Type: Observational
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Cemre Aydeğer, Reseach Asistant, Dr., Çanakkale Onsekiz Mart University
Other Study IDs: COMU-FNO-1
Record Dates: First submitted 2025-07-30; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-12

CONDITIONS: Oncology; Geriatric Oncology; Physiology
Keywords: geriatric oncology; chemotoxicity
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This prospective observational study aims to evaluate and compare the effectiveness of three geriatric assessment tools-CARG (Cancer and Aging Research Group score), G8 screening tool, and Frailty Scale-in predicting chemotherapy-related toxicity (CRT) in cancer patients aged 65 years and older. A total of at least 100 patients receiving standard chemotherapy (excluding hematologic malignancies and immunotherapy) at Çanakkale University Medical Faculty Oncology Clinic will be assessed prior to treatment initiation. Each participant will undergo baseline evaluations including G8, CARG, and Frailty assessments. The study will analyze the correlation between these tools and the occurrence of CRT using AUC, logistic regression, and correlation analyses. The goal is to identify the most accurate and practical screening tool to guide clinical decision-making and minimize chemotherapy toxicity in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older.
* Histologically confirmed cancer diagnosis with a pre-planned chemotherapy regimen (adjuvant, neoadjuvant, or palliative intent).
* Chemotherapy not yet initiated at the time of enrollment.
* Clinically stable condition, as assessed by the oncologist.
* Willingness and ability to provide written informed consent.

Exclusion Criteria:

* Presence of acute infection or advanced organ failure (cardiac, hepatic, or renal).
* Severe psychiatric illness or cognitive impairment that interferes with the ability to complete assessments.
* Patients receiving concurrent hormonal therapy, targeted therapy, immunotherapy, or radiotherapy.
* Diagnosis of hematologic malignancies (e.g., leukemia, lymphoma, myeloma).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will consist of adult oncology patients aged 65 years and older who are scheduled to receive systemic chemotherapy for solid tumors at the Çanakkale Onsekiz Mart University Medical Faculty, Department of Medical Oncology. Eligible participants must have a confirmed cancer diagnosis and a predefined chemotherapy regimen (adjuvant, neoadjuvant, or palliative), but must not have yet started treatment at the time of enrollment.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Geriartric Form Results and Chemotherapy Side Effects | From enrollment to 6 month
  ARG (Cancer and Aging Research Group score)
G8 screening tool | From enrollment to 6 month
  prediction side effets on chemotherapy on patient
Frailty Scale | From enrollment to 6 month
  Predicting side effect chemoterapy in elderly patient

CONTACTS AND LOCATIONS:
Locations (1):
- Çanakkale Onsekiz Mart Univercity, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Runzer-Colmenares FM, Urrunaga-Pastor D, Roca-Moscoso MA, De Noriega J, Rosas-Carrasco O, Parodi JF. Frailty and Vulnerability as Predictors of Chemotherapy Toxicity in Older Adults: A Longitudinal Study in Peru. J Nutr Health Aging. 2020;24(9):966-972. doi: 10.1007/s12603-020-1404-6. PMID 33155622
- [Background] Retornaz F, Guillem O, Rousseau F, Morvan F, Rinaldi Y, Nahon S, Castagna C, Boulahssass R, Grino M, Gholam D. Predicting Chemotherapy Toxicity and Death in Older Adults with Colon Cancer: Results of MOST Study. Oncologist. 2020 Jan;25(1):e85-e93. doi: 10.1634/theoncologist.2019-0241. Epub 2019 Aug 6. PMID 31387952
- [Background] Ostwal V, Ramaswamy A, Bhargava P, Hatkhambkar T, Swami R, Rastogi S, Mandavkar S, Ghosh J, Bajpai J, Gulia S, Srinivas S, Rath S, Gupta S. Cancer Aging Research Group (CARG) score in older adults undergoing curative intent chemotherapy: a prospective cohort study. BMJ Open. 2021 Jun 29;11(6):e047376. doi: 10.1136/bmjopen-2020-047376. PMID 34187825
- [Background] Kenis C, Bron D, Libert Y, Decoster L, Van Puyvelde K, Scalliet P, Cornette P, Pepersack T, Luce S, Langenaeken C, Rasschaert M, Allepaerts S, Van Rijswijk R, Milisen K, Flamaing J, Lobelle JP, Wildiers H. Relevance of a systematic geriatric screening and assessment in older patients with cancer: results of a prospective multicentric study. Ann Oncol. 2013 May;24(5):1306-12. doi: 10.1093/annonc/mds619. Epub 2013 Jan 4. PMID 23293115
- [Background] Juthani R, Punatar S, Mittra I. New light on chemotherapy toxicity and its prevention. BJC Rep. 2024 May 22;2(1):41. doi: 10.1038/s44276-024-00064-8. PMID 39516565
- [Background] Hurria A, Togawa K, Mohile SG, Owusu C, Klepin HD, Gross CP, Lichtman SM, Gajra A, Bhatia S, Katheria V, Klapper S, Hansen K, Ramani R, Lachs M, Wong FL, Tew WP. Predicting chemotherapy toxicity in older adults with cancer: a prospective multicenter study. J Clin Oncol. 2011 Sep 1;29(25):3457-65. doi: 10.1200/JCO.2011.34.7625. Epub 2011 Aug 1. PMID 21810685
- [Background] Goede V. Frailty and Cancer: Current Perspectives on Assessment and Monitoring. Clin Interv Aging. 2023 Mar 28;18:505-521. doi: 10.2147/CIA.S365494. eCollection 2023. PMID 37013130
- [Background] Feliu J, Jimenez-Munarriz B, Basterretxea L, Paredero I, Llabres E, Antonio-Rebollo M, Losada B, Espinosa E, Girones R, Custodio AB, Del Mar Munoz M, Diaz-Almiron M, Gomez-Mediavilla J, Pinto A, Torregrosa MD, Soler G, Cruz P, Higuera O, Molina-Garrido MJ. Predicting Chemotherapy Toxicity in Older Patients with Cancer: A Multicenter Prospective Study. Oncologist. 2020 Oct;25(10):e1516-e1524. doi: 10.1634/theoncologist.2019-0701. Epub 2020 Apr 30. PMID 32329131
- [Background] Decoster L, Van Puyvelde K, Mohile S, Wedding U, Basso U, Colloca G, Rostoft S, Overcash J, Wildiers H, Steer C, Kimmick G, Kanesvaran R, Luciani A, Terret C, Hurria A, Kenis C, Audisio R, Extermann M. Screening tools for multidimensional health problems warranting a geriatric assessment in older cancer patients: an update on SIOG recommendationsdagger. Ann Oncol. 2015 Feb;26(2):288-300. doi: 10.1093/annonc/mdu210. Epub 2014 Jun 16. PMID 24936581
- [Background] Church S, Rogers E, Rockwood K, Theou O. A scoping review of the Clinical Frailty Scale. BMC Geriatr. 2020 Oct 7;20(1):393. doi: 10.1186/s12877-020-01801-7. PMID 33028215
- [Background] Chon J, Timilshina N, AlMugbel F, Jin R, Monginot S, Tejero I, Breunis H, Alibhai SMH. Validity of a self-administered G8 screening test for older patients with cancer. J Geriatr Oncol. 2023 Sep;14(7):101553. doi: 10.1016/j.jgo.2023.101553. Epub 2023 Jun 26. PMID 37379768
- [Background] Bellera CA, Rainfray M, Mathoulin-Pelissier S, Mertens C, Delva F, Fonck M, Soubeyran PL. Screening older cancer patients: first evaluation of the G-8 geriatric screening tool. Ann Oncol. 2012 Aug;23(8):2166-2172. doi: 10.1093/annonc/mdr587. Epub 2012 Jan 16. PMID 22250183